CLINICAL TRIAL: NCT00144625
Title: An Open-label, Extension, Phase III Study to Evaluate the Long-term Safety, Efficacy and PK of MRA in Patients With pJIA Who Participated in Study MRA318JP
Brief Title: Long-term Treatment Study of MRA for Polyarticular Juvenile Idiopathic Arthritis (pJIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA319JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Polyarticular Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg/4weeks

SUMMARY:
This is an open-label, extension, Phase III study to evaluate the long-term safety, efficacy and PK of MRA in patients with pJIA who participated in Study MRA318JP.

ELIGIBILITY:
Inclusion criteria

* Of the patients who received three infusions with MRA in the previous study and for whom a last observation was conducted
* the patients who did not have problems with safety in the previous study"

Exclusion criteria

* Patients who were not enrolled by 3 months after completion of the previous study
* Patients who received any of the following since completion of the previous study until initiation of treatment in the present study

  1. DMARDs or immunosuppressants
  2. Intravenous and intramuscular injection of corticosteroids
  3. Plasma exchange therapy
  4. Other drugs and therapies that may affect evaluation of drug efficacy

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-02; Primary Completion 2005-07 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Efficacy:Percentage of patients showing 30% improvement in the JIA core set every 3M, LOBS | every 3 months
Safety:Incidence and severity of adverse events and adverse drug reactions | whole period
Pharmacokinetics:The time course of the trough values for the serum MRA concentration | whole period

SECONDARY OUTCOMES:
Efficacy:The time course of the percentage of patients showing 30%, 50%, and 70% improvement in the JIA core set, each variable of the JIA core set, CRP, pain every 3M, LOBS | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical